CLINICAL TRIAL: NCT07189156
Title: Immediate Versus Delayed Weight Bearing After Fixation of Pelvis and Acetabulum Fractures: A Multicenter Feasibility Randomized Controlled Trial
Brief Title: Weight Bearing After Pelvis and Acetabulum Fracture Fixation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, Peter Mittwede, Assistant Professor, University of Mississippi Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMMC-IRB-2025-115
Record Dates: First submitted 2025-08-26; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Pelvis Fractures; Acetabulum Fractures
Keywords: Weight Bearing; Pelvis Fractures; Acetabulum Fractures; Immediate Weight Bearing; Early Weight Bearing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient who has a pelvis fracture treated operatively (Experimental)
  Interventions: Other: Immediate Weight Bearing Pelvis; Other: Delayed Weight Bearing Pelvis
- Patient who has an acetabulum fracture treated operatively (Experimental)
  Interventions: Other: Immediate Weight Bearing Acetabulum; Other: Delayed Weight Bearing Acetabulum

INTERVENTIONS:
Other: Immediate Weight Bearing Pelvis — Patient with a pelvis fracture may be randomized to be immediately weight bearing as tolerated after surgery.
  Arms: Patient who has a pelvis fracture treated operatively
Other: Delayed Weight Bearing Pelvis — Patient with a pelvis fracture may be randomized to be delayed weight bearing as tolerated (either non-weight bearing, foot flat, or toe touch weight bearing per surgeon discretion) for 6-12 weeks after surgery.
  Arms: Patient who has a pelvis fracture treated operatively
Other: Immediate Weight Bearing Acetabulum — Patient with an acetabulum fracture may be randomized to be immediately weight bearing as tolerated after surgery.
  Arms: Patient who has an acetabulum fracture treated operatively
Other: Delayed Weight Bearing Acetabulum — Patient with an acetabulum fracture may be randomized to be delayed weight bearing as tolerated (either non-weight bearing, foot flat, or toe touch weight bearing per surgeon discretion) for 6-12 weeks after surgery.
  Arms: Patient who has an acetabulum fracture treated operatively

SUMMARY:
The goal of this study to determine if a randomized clinical trial of immediate versus delayed weight bearing after undergoing surgical fixation of a pelvis or acetabulum fracture is feasible. The main questions it aims to answer are:

Are surgeons willing to allow inclusion of their patients into such a trial? Are patients willing to participate in such a trial? Will patients be compliant with assigned weight bearing status in such a trial? Can good patient follow-up be obtained in such a trial? Is participation in such a trial safe?

Patients from 7 medical centers will be enrolled, and randomized to immediate weight bearing as tolerated (WBAT) versus delayed WBAT (for 6-12 weeks). Feasibility metrics revolving around enrollment, follow-up, and documentation will be monitored, as well as medical and surgical complications. This pilot study will help inform feasibility and design of a larger definitive multicenter randomized controlled trial (RCT) on this topic.

DETAILED DESCRIPTION:
Early weight bearing is frequently allowed and encouraged following fixation of hip and femoral and tibial shaft fractures, while periarticular and pelvis and acetabulum fractures are often prescribed 6-12 weeks of restricted weight bearing. Early weight bearing has been shown to be associated with a number of benefits following fixation of various lower extremity fractures, and delayed weight bearing is associated with an increased risk of medical complications and delayed improvement in functional outcomes. The risks associated with delayed weight bearing have encouraged clinicians to consider the safety of early weight bearing after fixation of various lower extremity fractures.

Retrospective studies have shown low rates of hardware failure with early weight bearing following fixation of fractures for which early WBAT has not traditionally been allowed, including fractures of the pelvis, acetabulum, distal femur, proximal tibia, and distal tibia. Randomized controlled trials with ankle and distal femur fractures have shown no difference in rates of early hardware failure between early and delayed weight bearing. However, high-quality studies in pelvis and acetabulum are lacking.

A definitive RCT on early versus delayed WBAT after fixation of pelvis and acetabulum fractures is necessary, and this would focus on important outcomes such as surgical and medical complications, patient-reported functional status, and timing of return to work or activities of daily living. However, a pilot trial of adequate size is needed to highlight 1) if participant enrollment is feasible (from a surgeon and patient perspective), and 2) if appropriate follow-up and compliance with documentation can be achieved. A pilot trial would also help establish the safety of such a trial, as perioperative complications would be monitored.

The completion of this pilot trial will assist with the design and implementation of a definitive RCT that will compare patient-relevant outcomes of immediate versus delayed WBAT following fixation of pelvis and acetabulum fractures.

RESEARCH QUESTION Is a randomized controlled trial (RCT) of immediate versus delayed weight bearing following fixation of fractures of the pelvis and acetabulum feasible?

SCIENTIFIC AIMS The proposed feasibility trial will address the paucity of high-quality data regarding the safety and feasibility of early weight bearing following fixation of pelvis and acetabulum fractures. A high amount of variability exists with these fractures with regard to the severity of bony, soft tissue, and non-orthopaedic injuries, so our feasibility criteria include: 1) 25% overall patient enrollment (with surgeon and patient agreement to participate in 50% of eligible cases each), 2) >90% follow-up at 3 months), 3) 100% correct documentation of weight bearing status, and 4) 100% correct documentation of primary outcome of reoperation.

HYPOTHESIS The investigators hypothesize that the feasibility criteria will be met, and that this pilot study will inform the design and implementation of a definitive RCT on this topic.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 years old and above
2. Patients with surgically treated pelvis or acetabulum fractures

Exclusion Criteria:

1. Presence of fractures to the ipsilateral or contralateral lower extremity that would preclude WBAT on the surgically repaired pelvis/acetabulum fracture
2. Presence of upper extremity injury that would limit weight bearing using an assistive device such as a walker or crutches
3. Severe injuries to other body systems that would prevent patient from being able to comply with weight bearing protocol
4. Presence of significant psychiatric or cognitive disorder or disability that would prevent patient from being able to comply with weight bearing protocol
5. Pre-injury non-ambulatory status
6. Suspected issues with follow-up
7. Language barriers precluding obtaining adequate informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Study enrollment rates of eligible patients | Within 72 hours after surgery
  Target enrollment of 50% of patients (surgeon agreement to enroll patient) and 50% of patients eligible for inclusion to agree to participate in study
Clinic follow-up rates for patients enrolled in study | 3 months
  >90% target follow-up of patients at 3-month postoperative visit
Correct documentation of randomized weight bearing status in medical charts of patients | 12 months
  Target 100% correct documentation of assigned weight bearing status in postoperative medical documentation (both in-hospital documentation and during follow-up visits)
Correct documentation of secondary outcome of reoperation in medical documentation | 12 months
  Target 100% correct documentation of secondary outcome of reoperation in medical documentation during follow-up visits

SECONDARY OUTCOMES:
Patient reoperation for any reason in the postoperative period | 12 months
  Track number of all-cause reoperations in all patients in medical documentation postoperatively

CONTACTS AND LOCATIONS:
Locations (7):
- United States (6):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Arrowhead Regional Medical Center, Colton, California
  - Indiana University Health, Indianapolis, Indiana
  - R Adams Cowley Shock Trauma Center - University of Maryland, Baltimore, Maryland
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Inova Medical Group, Fairfax, Virginia
- Vancouver General Hospital - University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided